CLINICAL TRIAL: NCT05528055
Title: A Phase I Study to Investigate the Safety, Tolerability, Preliminary Efficacy and Pharmacokinetics(PK) of SCR-6920 Capsule in Patients With Advanced Malignant Tumors
Brief Title: A Study to Investigate the Safety and Tolerability of SCR-6920 Capsule in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM1907-04-PRMT5-101
Record Dates: First submitted 2022-05-10; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumor; Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose escalation (Experimental): Participants will receive SCR-6920 capsule orally at escalating doses, till the maximum tolerated dose level is reached, and the recommended phase 2 dose(RP2D) will be determined.
  Interventions: Drug: SCR-6920 capsule
- Dose expansion: non small cell lung cancer(NSCLC) (Experimental): Participants will receive SCR-6920 capsule orally at the recommended phase 2 dose
  Interventions: Drug: SCR-6920 capsule
- Dose expansion: NHL (Experimental): Participants will receive SCR-6920 capsule orally at the recommended phase 2 dose on a continuous basis
  Interventions: Drug: SCR-6920 capsule
- Dose expansion: solid tumors (Experimental): Participants will receive SCR-6920 capsule orally at the recommended phase 2 dose on a continuous basis
  Interventions: Drug: SCR-6920 capsule

INTERVENTIONS:
Drug: SCR-6920 capsule — SCR-6920 capsule will be oral administered once daily at escalating doses on a continuous basis
  Other Names: PRMT5 inhibitor
  Arms: Dose escalation
Drug: SCR-6920 capsule — SCR-6920 capsule will be oral administered once daily at the recommended phase 2 dose on a continuous basis
  Other Names: PRMT5 inhibitor
  Arms: Dose expansion: non small cell lung cancer(NSCLC)
Drug: SCR-6920 capsule — SCR-6920 capsule will be oral administered once daily at the recommended phase 2 dose on a continuous basis
  Other Names: PRMT5 inhibitor
  Arms: Dose expansion: NHL
Drug: SCR-6920 capsule — SCR-6920 capsule will be oral administered once daily at the recommended phase 2 dose on a continuous basis
  Other Names: PRMT5 inhibitor
  Arms: Dose expansion: solid tumors

SUMMARY:
A Phase 1, open label, multi center, dose escalation and expansion study will assess the safety, tolerability, PK, and preliminary efficacy of SCR-6920 capsule in participants with advanced malignant tumors. The purpose of the study is to identify the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D), and to confirm the tolerability and preliminary efficacy of SCR-6920 in participants with advanced solid tumors and relapsed/refractory non-Hodgkin lymphoma(NHL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumors or histopathologically confirmed NHL
* Relapsed/refractory solid tumor or relapsed/refractory NHL who have progressed during or after standard therapy or for which treatment is not tolerated, not suitable, not available.
* At least one evaluable or measurable lesion (as defined in the protocol).
* ECOG Performance Status 0 or 1.
* Life expectancy ≥12 weeks.
* Adequate organ function (as defined in the protocol).
* Reproductive criteria (as defined in the protocol).

Exclusion Criteria:

* Any clinically significant gastrointestinal (GI) abnormalities that may alter absorption.
* Major surgery, systemic anti-cancer therapy or investigational drug(s) within 4 weeks prior to study entry. Radiation therapy within 2 weeks prior to study entry.
* Adverse reactions from previous anti-tumor therapy have not yet recovered to ≤ grade 1(excluding hair loss, peripheral neurotoxicity caused by chemotherapy have recovered to ≤ grade 2 ).
* Autologous hematopoietic stem cell transplantation was performed within 9 months prior to the first dose.
* History of a second malignancy within 2 years (as defined in the protocol).
* Active uncontrolled or symptomatic lung disease (as defined in the protocol).
* Intracranial hypertension or active uncontrolled or symptomatic CNS metastases.
* Known or suspected hypersensitivity to study medications.
* Known active uncontrolled or symptomatic CNS metastases.
* The investigator determined that the patient should not participate in the study.
* Known mental illness or substance abuse that may disrupt therapy.
* Clinically significant cardiac abnormalities (as defined in the protocol).
* Gestating or Lactating women.
* Pleural effusion, pericardial effusion or ascites that need diuretics or draining within 2 weeks prior to first dose.
* The patient is currently using a drug known to be a strong inhibitor or inducer of CYP3A4.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity(DLT) | Up to 28 days
  DLT will be evaluated within 28 days since first dose. The number of DLTs will be used to determine the maximum tolerated dose (MTD).
Overall Response Rate (ORR) | Up to approximately 1 years
  Participants with solid tumor: ORR based on RECIST1.1 criteria; Participants with NHL: ORR based on Lugano criteria

SECONDARY OUTCOMES:
Number of participants with any adverse events (AEs), serious adverse events (SAEs), withdrawal due to AEs, dose interruptions and reductions | Up to approximately 1 years
  All AEs, SAEs and dose modifications will be collected. Adverse events as characterized by type, severity, timing and relationship to study therapy. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Number of participants with clinically significant changes in laboratory parameters, vital signs, electrocardiogram (ECG), physical examination and organ-specific parameters. | Up to approximately 1 years
  Blood and urine samples will be collected for analysis of lab parameters. Vital signs, electrocardiogram (ECG), physical examinations and organ-specific parameters will be collected at specified time points. Number of participants with clinically significant changes in laboratory parameters, vital signs, electrocardiogram (ECG), physical examination and organ-specific parameters will be reported.
Pharmacokinetic Parameters: Area Under the Curve (AUC) | Up to approximately 1 years
  Blood samples will be collected at given time points to determine the AUC (0-t) and AUC (0-inf) of SCR-6920
Pharmacokinetic Parameters: Maximum Concentration (Cmax) | Up to approximately 1 years
  Blood samples will be collected at given time points to determine the Cmax of SCR-6920.
Pharmacokinetic Parameters: Trough Concentration (Ctrough) | Up to approximately 1 years
  Blood samples will be collected at given time points to determine the Ctrough of SCR-6920.
Pharmacokinetic Parameters: Time to Maximum Concentration (Tmax) | Up to approximately 1 years
  Blood samples will be collected at given time points to determine the Tmax of SCR-6920.
Pharmacokinetic Parameters: Terminal elimination half life (t1/2) | Up to approximately 1 years
  Blood samples will be collected at given time points to determine the t1/2 of SCR-6920.
Change from Baseline in symmetrical arginine dimethylation (SDMA) as a PD measure | Up to approximately 1 years
  Evaluation of change from baseline in SDMA, a PD biomarker of PRMT5 inhibition.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China